CLINICAL TRIAL: NCT06319651
Title: Effects of Lower Limb Resistance Band Exercises in Phase 1 Cardiac Rehabilitation on Functional Recovery Among Post Coronary Artery Bypass Grafting Patients
Brief Title: Effects of Lower Limb Resistance Band Exercises in Phase 1 Cardiac Rehabilitation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: REC/RCR&AHS/23/0360
Record Dates: First submitted 2024-03-04; First posted 2024-03-20 (Actual); Last update posted 2024-07-23 (Actual); Status verified 2024-07

CONDITIONS: Cardiovascular Diseases
Keywords: Coronary artery bypass grafting; Cardiac rehabilitation; Resistance band exercise
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial (RCT). Pre & Post data collection
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): In addition to the routine Phase 1 cardiac rehabilitation, Resistance Exercises
  * Extending thighs
  * Closing thighs
  * Opening thighs
  * Bending thighs
  * Bending ankles
  * Ankle opening
  Interventions: Other: Lower Limb Resistance Band Exercises; Other: Routine Phase 1 cardiac rehabilitation
- Routine Phase 1 cardiac rehabilitation (Active Comparator): Routine Phase 1 cardiac rehabilitation only.
  Interventions: Other: Routine Phase 1 cardiac rehabilitation

INTERVENTIONS:
Other: Lower Limb Resistance Band Exercises — * Extending thighs
  * Closing thighs
  * Opening thighs
  * Bending thighs
  * Bending ankles
  * Ankle opening
  Arms: Experimental Group
Other: Routine Phase 1 cardiac rehabilitation — Routine Phase 1 cardiac rehabilitation only.

SUMMARY:
This study will be randomized controlled trial with non-probability purposive sampling. Study conducted among post CABG patients. Sample size will be 56, 28 in each group. Outcome will be measured by using 6 minute walk test, Spirometry (FVC, FEV1/FVC and PEF), Functional Independence Measure.

DETAILED DESCRIPTION:
This study will be randomized controlled trial with non-probability purposive sampling. Study conducted among post CABG patients. Descriptive analysis will be applied. Data will be collected from Rehmatul lil Alameen Institute of cardiology Lahore. Sample size will be 56, 28 in each group. In addition to the routine Phase 1 cardiac rehabilitation for experimental group the exercise protocol consisted of 10 minutes of warm up, elastic band strength exercise protocol (30 minutes) and cool down (5 minutes) so that an exercise session lasted about 45-50 minutes, exercise will performed circularly 2 sets, 10 repetition with a 2 minute rest after each cycle and monitored the performance of exercise for 6 days. Resisted band exercise are Extending thighs, Closing thighs, Opening thighs, Bending thighs, Dorsiflexion, Plantarflexion. For control group routine Phase 1 cardiac rehabilitation only. Outcome will be measured by using 6 minute walk test, Spirometry (FVC, FEV1/FVC and PEF), Functional Independence Measure.

ELIGIBILITY:
Inclusion Criteria:

* Age 35 to 60
* Female and Male both
* Hemodynamic stable patients
* Arrhythmias or angina not present
* Post elective sternotomy surgery
* Post extubating

Exclusion Criteria:

* Chronic obstructive pulmonary disease
* Neurological Sequelae
* Neuromuscular disease
* Emergency or off pump surgery
* Surgical re-intervention
* Patient who remained on mechanical ventilation longer than 24 hours
* Patient who had a baseline partial pressure of oxygen (PaO2) less than 75 mmHg and partial pressure of carbon dioxide (PCO2) 45 mmHg
* Patients who had history of respiratory tract infection within a period of three months

Ages: 35 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2024-03-01 (Actual); Primary Completion 2024-06-05 (Actual); Study Completion 2024-06-15 (Actual)

PRIMARY OUTCOMES:
Functional Independence Measure | 6 Days
  The Functional Independence Measure (FIM) is an instrument that was developed as a measure of disability for a variety of populations and is not specific to any diagnosis. The FIM instrument Includes measures of independence for self-care, including sphincter control, transfers, locomotion, communication, and social cognition.
  Is an 18-item, seven-level, ordinal scale intended to be sensitive to changes over the course of a comprehensive inpatient medical rehabilitation program.
  Uses the level of assistance an individual needs to grade functional status from total independence to total assistance).
  The tool is used to assess a patient's level of disability as well as a change in patient status in response to rehabilitation or medical intervention.
  FIM 3 levels.
6 Minute Walk Test | 6 Days
  The 6 Minute Walk Test is a sub-maximal exercise test used to assess aerobic capacity and endurance. The distance covered over a time of 6 minutes is used as the outcome by which to compare changes in performance capacity
Forced expiratory volume (FEV1) | 6 Days
  Forced expiratory volume (FEV1) calculates the amount of air that a person can force out of their lungs in 1 second. It's measured by spirometry
Forced vital capacity (FVC) | 6 Days
  Forced vital capacity (FVC) is the amount of air that can be forcibly exhaled from your lungs after taking the deepest breath possible. It's measured by spirometry
FEV1/FVC ratio | 6 Days
  The FEV1/FVC ratio is the ratio of the forced expiratory volume in the first one second to the forced vital capacity of the lungs. The normal value for this ratio is above 0.75-85. It's measured by spirometry

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Faizan Hamid, Ms-CPPT, Principal Investigator — Riphah International University
Locations (1):
- Rehmatul lil Alameen Institute of cardiology, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No